CLINICAL TRIAL: NCT03864328
Title: Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Efficacy and Safety Study With Inhaled RVT-1601 for the Treatment of Persistent Cough in Patients With Idiopathic Pulmonary Fibrosis (IPF): SCENIC Trial
Brief Title: A Phase 2b Study of Inhaled RVT-1601 for the Treatment of Persistent Cough in IPF
Acronym: SCENIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: Respivant Sciences GmbH (Industry)
Collaborators: Respivant Sciences Inc. (Industry)
Responsible Party: Sponsor
Organization: Respivant Sciences Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT1601-CC-04
Record Dates: First submitted 2019-03-02; First posted 2019-03-06 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Persistent Cough in IPF; Chronic Cough; IPF
Keywords: Cough; Chronic Cough; IPF; IPF Cough
MeSH Terms: conditions — Chronic Cough; Cough

STUDY DESIGN:
Intervention Model Description: Randomization stratified by background IPF therapy use and FVC % predicted at baseline
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RVT-1601 Low Dose (Experimental)
  Interventions: Drug: RVT-1601
- RVT-1601 Mid Dose (Experimental)
  Interventions: Drug: RVT-1601
- RVT-1601 High Dose (Experimental)
  Interventions: Drug: RVT-1601
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RVT-1601 — Inhaled RVT-1601 administered TID via eFlow nebulizer
  Arms: RVT-1601 High Dose; RVT-1601 Low Dose; RVT-1601 Mid Dose
Drug: Placebo — Inhaled Placebo administered TID via eFlow nebulizer
  Arms: Placebo

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a rare, progressive life-threatening disease that is characterized by exertional dyspnea and persistent dry cough.

Cough in IPF is both a presenting and a complicating clinical feature, which affects approximately three quarters of IPF cases. It is often a debilitating symptom that adversely affects quality of life (QoL) and is usually refractory to medical therapy.

Inhaled RVT-1601 (formerly, PA101B), a new inhalation formulation of cromolyn sodium delivered via the eFlow® Closed System (CS) nebulizer, is being evaluated in this Phase 2b study for the treatment of persistent cough in patients with IPF.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 40 through 89 years
* Confirmed diagnosis of IPF with clinical features consistent with the current clinical practice guidelines
* Persistent cough for at least 8 weeks that is primarily due to IPF and not responsive to anti-tussive therapy
* Daytime cough severity score of ≥ 40 mm on a 100-mm VAS
* 24-hour average cough count of at least 10 coughs per hour
* Forced Vital Capacity (FVC) > 45% predicted value within 4 weeks
* Diffusion capacity for carbon monoxide corrected for hemoglobin (DLCOc) > 30% predicted value within 4 weeks
* Life expectancy of at least 12 months

Exclusion Criteria:

* Current or recent history of clinically significant medical condition, laboratory abnormality, or illness that could place the subject at risk or compromise the quality of the study data
* Significant coronary artery disease (i.e., myocardial infarction within 6 months or unstable angina within 1 month)
* Upper or lower respiratory tract infection within 4 weeks
* Acute exacerbation of IPF within 6 months
* Lung transplantation expected within 12 months
* Requiring supplemental O2 > 4 litres/min to maintain peripheral arterial O2 saturation (SpO2) > 88% at rest
* History of malignancy likely to result in significant disability or likely to require significant medical or surgical intervention within the next 2 years
* Current smoker (i.e., use of tobacco products within the last 3 months)
* Current or recent history of drug or alcohol abuse within 12 months
* Participation in any other investigational drug study within 4 weeks
* Use of certain drugs for cough management within 4 weeks: prednisone, opiates, baclofen, gabapentin, pregabalin, thalidomide, amitriptyline, inhaled corticosteroids, or inhaled bronchodilators
* Use of ACE inhibitors or cromolyn sodium within 4 weeks
* Females who are pregnant or breastfeeding, or if of child-bearing potential unwilling to practice acceptable means of birth control during the study
* History of hypersensitivity or intolerance to cromolyn sodium

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour average cough count | 12 weeks
  Objective cough count monitoring performed using a digital recording device.

SECONDARY OUTCOMES:
Change in cough severity | 12 weeks
  Cough severity assessed using Visual Analog Scale (VAS), a single-item questionnaire using 100-point scale ranging from 0 (no cough) to 100 (extremely severe cough).
Change in cough-specific QoL | 12 weeks
  Cough-specific QoL assessed using Leicester Cough Questionnaire (LCQ), a 19-item questionnaire designed to measure impact of cough in three domains (physical, psychological and social), each domain ranging from 1 to 7 and LCQ total score ranging from 3 to 21, with the higher scores corresponding with better QoL.

OTHER OUTCOMES:
Change in forced vital capacity (FVC) | 12 weeks
  FVC measured as the total amount of air exhaled during pulmonary function test.
Change in disease-specific QoL | 12 weeks
  Disease-specific QoL assessed using King's Brief Interstitial Lung Disease Questionnaire (K-BILD), a 15-item questionnaire designed to measure impact of interstitial lung disease in three domains (breathlessness and activities, psychological and chest symptoms), each domain and total score ranging from 0 to 100 with the higher scores corresponding with better QoL.
Change in airway and lung volumes as measured by HRCT images | 12 weeks
  HRCT-based functional respiratory imaging (FRI) parameters measured at end-inspiration and end-expiration.
Change in biomarkers | 12 weeks
  Collagen degradation by-products measured in the blood.
Change in respiratory-related QoL | 12 weeks
  Respiratory-related QoL assessed using St. George's Respiratory Questionnaire (SGRQ), a 50-item questionnaire designed to measure impact of respiratory symptoms on overall health, daily life, and perceived well-being, with total score ranging from 0 to 100 and lower score denoting a better health status.
Change in dyspnea score | 12 weeks
  Dyspnea score assessed using University of California San Diego (UCSD) Shortness of Breath Questionnaire (SOBQ),a 24-item questionnaire designed to measure breathlessness on a scale from 0 (not at all breathless) to 5 (maximally breathless or too breathless to do the activity).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Tutuncu, MD, PhD, Study Director — Respivant Sciences Inc.
Locations (81):
- United States (28):
  - University of Alabama, Birmingham, Alabama
  - University of California Davis, Sacramento, California
  - University California San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Ascension Medical Group / St. Vincent's Lung Institute, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Tampa General Hospital / Uni of South Florida, Tampa, Florida
  - Loyola University, Maywood, Illinois
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Universty of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - Cornell University Weill Cornell Medical College, New York, New York
  - American Health Research, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Pulmonix, LLC, Greensboro, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwester Medical Center, Dallas, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington School of Medicine, Seattle, Washington
- Australia (10):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Lung Research Quensland, Chermside, Quensland
  - Mater Research, South Brisbane, Quensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Frankston Hospital-Peninsula Health, Frankston, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Health, Westmead, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Trialswest, Perth, Western Australia
- Belgium (2):
  - University Clinic Saint-Luc, Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
- Canada (5):
  - Dalhousie University, Halifax
  - McMaster University, Hamilton
  - Centre Hospitalier Universitaire de Montreal, Montreal
  - University Health Network, Toronto General Hospital, Toronto
  - St. Paul's Hospital, Vancouver
- Thomayer Hospital, Prague, Czechia
- Germany (8):
  - Evangelische Lungerklinik Berlin, Berlin
  - University Clinic Bonn, Bonn
  - Ruhrlandklinik-Universitätsmedizin Essen, Essen
  - Pneumologische Klinik Waldhof Elgerhausen, Greifenstein
  - Medizinische Hochshule Hannover, Hanover
  - University Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Krankenhaus Bethanian, Solingen
- Italy (7):
  - Bologna University Hospital, Bologna
  - University of Catania, Catania
  - A.O.U. Policlinico di Modena, Modena
  - University of Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Siena University Hospital, Siena
  - University of Torino, Torino
- Netherlands (5):
  - VU Medical Center, Amsterdam
  - Zuyderland Medical Center, Heerlen
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medical Center, Rotterdam
  - Haaglanden Medical Center, The Hague
- New Zealand (3):
  - Greenlane Clinical Center, Auckland
  - University of Otago, Christchurch
  - Waikato Hospital, Hamilton
- Turkey (Türkiye) (3):
  - Cukurova University, Adana
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Ege University Hospital, Izmir
- United Kingdom (9):
  - Castle Hill Hospital, Cottingham, East Yorkshire
  - Royal Papworth Hospital, Cambridge
  - University of Edinburgh, Edinburgh
  - University of Leicester, Leicester
  - University Hospital Aintree, Liverpool
  - Royal Brompton Hospital, London
  - University of Manchester, Manchester
  - Nottingham University Hospital, Nottingham
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No